CLINICAL TRIAL: NCT04476108
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY3016859 for the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: Chronic Pain Master Protocol (CPMP): A Study of LY3016859 in Participants With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17535; H0P-MC-NP01 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 750 Mg-500 mg LY3016859 (Experimental): Participants received LY3016859 every 2 weeks with 750 mg as starting dose followed by 500 mg intravenous (IV) infusion for a total of 4 doses.
  Interventions: Drug: LY3016859
- Placebo (Placebo Comparator): Participants received LY3016859 every 2 weeks with 750 mg as starting dose followed by 500 mg IV infusion for a total of 4 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3016859 — Administered IV
  Arms: 750 Mg-500 mg LY3016859
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
This study is being done to test the safety and efficacy of the study drug LY3016859 for the treatment of diabetic peripheral neuropathic pain. This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a value of ≤30 on the pain catastrophizing scale.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions for the duration of the study.
* Have daily symmetrical foot pain secondary to peripheral neuropathy present for at least 6 months and as diagnosed through use of the Michigan Neuropathy Screening Instrument Part B ≥3 (©University of Michigan).
* Have a history and current diagnosis of type 1 or type 2 diabetes mellitus.
* Have stable glycemic control as indicated by a glycated hemoglobin ≤11 at time of screening.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have second- or third-degree atrioventricular (AV) heart block or AV dissociation or history of ventricular tachycardia.
* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* There is an inability to rule out other causative or confounding sources of pain in the primary condition under study.
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have congenital QT prolongation or QT interval corrected for heart rate using Fridericia's formula (QTcF) interval measurement >450 milliseconds (msec) for male participants, >470 msec for female participants, or >480 msec for participants with bundle branch block.
* Have any clinically important abnormality at screening, as determined by investigator, in physical or neurological examination, vital signs, electrocardiogram (ECG), or clinical laboratory test results that could be detrimental to the participant or could compromise the study.
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Have a current drug-induced neuropathy, for example, due to some types of chemotherapy, or other types of peripheral neuropathy.
* Have known hereditary motor, sensory or autonomic neuropathies.
* Have an estimated glomerular filtration rate (eGFR) of less than 70 milliliters/minute/1.73m² during screening.
* Have any clinically serious or unstable cardiovascular, musculoskeletal disorder, gastrointestinal, endocrinologic, hematologic, hepatic, metabolic, urologic, pulmonary, dermatologic, immunologic, or ophthalmologic disease within 3 months of baseline.
* Have megaloblastic anemia or combined degeneration of the spinal cord.
* Have received any antibodies against nerve growth factor (NGF), or antibodies against EGFR, or EGFR tyrosine kinase inhibitors.
* Have a history of allergic reactions to monoclonal antibodies, or clinically significant multiple or severe drug allergies, including but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis.
* Have a history or presence of uncontrolled asthma, eczema, significant atopy, significant hereditary angio-edema or common variable immune deficiency.
* Have fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (35):
  - Simon Williamson Clinic, Birmingham, Alabama
  - Synexus - US, Chandler, Arizona
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Irvine Clinical Research Center, Irvine, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Suncoast Research Group, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus - US, Orlando, Florida
  - Synexus - US, Pinellas Park, Florida
  - Martin E. Hale M.D., P.A., Plantation, Florida
  - Synexus Clinical Research US, Inc - Orlando, The Villages, Florida
  - Synexus Clinical Research, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Cotton O'Neil Infusion Center, Topeka, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Synexus - US, Omaha, Nebraska
  - PharmQuest, Greensboro, North Carolina
  - Synexus - Cincinnati, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Synexus - US, Dallas, Texas
  - Synexus - US, San Antonio, Texas
  - Synexus - US, Murray, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Latin Clinical Trial Center, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] James DE, Bailey J, van der Walt JS, Winkler J, Schoemaker R. Population Pharmacokinetics and Pharmacodynamics of Fepixnebart (LY3016859) and Epiregulin in Patients with Chronic Pain. Clin Pharmacokinet. 2025 May;64(5):757-767. doi: 10.1007/s40262-025-01506-3. Epub 2025 Apr 23. PMID 40266472
- See also: A Study of LY3016859 in Participants With Diabetic Peripheral Neuropathic Pain — https://trials.lillytrialguide.com/en-US/trial/56qE3cITLpaXlG6KcqLoKQ

RESULTS

PARTICIPANT FLOW:
Groups:
- 750 Mg-500 Milligram (mg) LY3016859: Participants received LY3016859 every 2 weeks with 750 mg as starting dose followed by 500 mg IV infusion for a total of 4 doses.
- Placebo: Participants received placebo every 2 weeks by IV infusion for a total of 4 doses.
Period: Overall Study
Arm/Group | 750 Mg-500 Milligram (mg) LY3016859 | Placebo
Started | 84 | 41
Received at Least 1 Dose of Study Drug | 83 | 41
Completed | 76 | 38
Not Completed | 8 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Inadvertent Enrollment | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 750 Mg-500 mg LY3016859: Participants received LY3016859 every 2 weeks with 750 mg as starting dose followed by 500 mg IV infusion for a total of 4 doses.
- Total: Total of all reporting groups
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo | Total
Number analyzed (Participants) | 84 | 41 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 24 | 74
  >=65 years | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.5) | 63.3 (8.9) | 62.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 14 | 49
  Male | 49 | 27 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 4 | 16
  White | 68 | 33 | 101
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84 | 41 | 125
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  score on a scale | 5.97 (1.69) | 6.30 (1.62) | 6.08 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the NRS
Description: The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95% credible interval (CrI) was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: All enrolled or randomized participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 70 | 38
score on a scale | -1.98 [-2.42 to -1.55] | -1.56 [-2.17 to -0.96]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = -0.42, 95% CI 2-sided [-1.17 to 0.32] — The Bayesian analyses include posterior probabilities instead of p-values, and 95% credible intervals instead of 95% confidence intervals

2. Secondary Outcome: Change From Baseline in the Brief Pain Inventory-Short Form (BPI-SF) Total Interference Score
Description: The BPI-SF is a numeric rating scale that assesses the severity of pain (severity scale), its impact on daily functioning (Interference scale), and other aspects of pain (for example, location of pain, relief from medications) in various disease states. BPI-SF score ranges from 0 = no pain to 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 75 | 38
score on a scale | -2.11 [-2.55 to -1.65] | -1.74 [-2.35 to -1.12]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = -0.37, 95% CI 2-sided [-1.09 to 0.35] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of Change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1 = very much better, and 7 = very much worse.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 76 | 38
score on a scale | 2.48 [2.25 to 2.72] | 2.75 [2.41 to 3.09]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = -0.27, 95% CI 2-sided [-0.69 to 0.15] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 70 | 38
score on a scale | -2.10 [-2.54 to -1.66] | -1.66 [-2.27 to -1.04]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = -0.44, 95% CI 2-sided [-1.20 to 0.31] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0 = no pain, and 100 = worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 76 | 38
score on a scale | -26.17 [-31.48 to -20.84] | -23.31 [-30.80 to -15.88]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = -2.86, 95% CI 2-sided [-11.71 to 6.06] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline Assessment to Endpoint on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale)
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Participants reported how often each sleep symptom or problem was present on a 5-point categorical scale ranging from 'all of the time' to 'none of the time.' It includes 12 questions with the first question assessing how long it takes the subject to fall asleep. The second question asks how many hours each night the subject slept. The remaining 10 questions have a range of 6 responses from 1="all of the time" to 6="none of the time". MOS Sleep scale scores range from 0 (min) to 100 (max). The original survey items are converted to a 0 to 100 range (by Converting 1 to 0, 2 to 25, 3 to 50, 4 to 75, and 5 to 100). Higher scores represent worse outcomes.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian longitudinal model.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 76 | 38
score on a scale | 0.21 [-0.05 to 0.47] | -0.14 [-0.51 to 0.22]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = 0.35, 95% CI 2-sided [-0.09 to 0.78] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Dosage Per Week
Description: Total Amount of Rescue Medication Use as Measured by Average Dosage per Week. Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg per week
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 70 | 38
mg per week | 271.58 [162.12 to 381.44] | 271.24 [118.00 to 426.01]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = 0.34, 95% CI 2-sided [-188.46 to 187.97] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline on the EuroQol-5D 5 Level Questionnaire (EQ-5D-5L) (United States)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than death) with higher scores indicating better health: 0 = a health state equivalent to death, and 1 = perfect health.
  Posterior mean change from baseline, 95% CrI was derived using Bayesian mixed model repeated measures.
Time Frame: Baseline, up to Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
Number analyzed (Participants) | 76 | 38
score on a scale | 0.07 [0.03 to 0.11] | 0.03 [-0.02 to 0.08]
Statistical Analysis 1: Comparison: 750 Mg-500 mg LY3016859 vs Placebo; Test type: Superiority; Bayesian Mixed Model Analysis; Posterior Mean Difference = 0.04, 95% CI 2-sided [-0.01 to 0.10] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through Week 26
Description: All enrolled or randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 750 Mg-500 mg LY3016859 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/83 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/83 | 2/41
Other Adverse Events (participants affected / at risk) | 28/83 | 12/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 750 Mg-500 mg LY3016859 (N=83) | Placebo (N=41)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 750 Mg-500 mg LY3016859 (N=83) | Placebo (N=41)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Infusion site pain (General disorders) | 4 (4) | 0 (0)
Xerosis (General disorders) | 3 (3) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT04476108/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04476108/SAP_001.pdf